CLINICAL TRIAL: NCT00175786
Title: Neuroradiologic Screening of Patients With Normal Tension Glaucoma
Brief Title: Magnetic Resonance Imaging of Patients With Normal Tension Glaucoma
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Frederick Mikelberg, University of British Columbia
Other Study IDs: C04-0404
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Normal Tension Glaucoma
Keywords: Glaucoma; Normal Tensions Glaucoma; Neuroradiology; Tumor; MRI; Magnetic Resonance Imaging; Compressive Lesion
MeSH Terms: conditions — Low Tension Glaucoma; Glaucoma; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to study the occurrence rate of masses such as brain tumors in patients with newly diagnosed Normal Tension Glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Lack of understanding of the study
* Unable or unwilling to undergo MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Mikelberg, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver Hospital and Health Sciences Centre, Vancouver, British Columbia, Canada